CLINICAL TRIAL: NCT07048977
Title: Comparison of Early Needle-knife Precut Papillotomy Over a Pancreatic Stent and Transpancreatic Sphincterotomy in Difficult Cannulation: A Prospective Randomized Controlled Trial
Brief Title: Early NK Precut vs TPS in Difficult Cannulation: A RCT (ENKPT Trial)
Acronym: ENKPT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Liang Chih-Ming, Deputy Director of Division of Hepato-Gastroenterology, Clinical Associate Professor., Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB 202101221A3; IRB 202101221A3 (Other: Kaohsiung Chang Gung Memorial Hospital)
Record Dates: First submitted 2025-06-17; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: ERCP Surgery
Keywords: Early Needle-knife Precut Papillotomy; Transpancreatic Sphincterotomy; Difficult Cannulation

STUDY DESIGN:
Intervention Model Description: The "difficult CBD cannulation" was defined as unsuccessful CBD cannulation after 5 minutes (stopwatch count) or three passes of the guidewire into the MPD. If the patients with three passes of the guidewire into the MPD were randomly assigned, in a 1:1 ratio, to needle knife precut papillotomy following the pancreas stent placement (NKP-SIPS group) or tranpancreatic sphincterotomy followed by the pancreas stent placement (TPS group ).
Who Masked: Participant
Masking Description: Patients are randomized into two groups at the time of providing informed consent by a 1:1 ratio, by opening a sealed envelope containing a noted marked with both groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NKP-SIPS group (Experimental): knife precut papillotomy following the pancreas stent placement
  Interventions: Procedure: Needle-Knife Precut Papillotomy over Pancreatic Stent
- TPS group (Active Comparator): Tranpancreatic sphincterotomy followed by the pancreas stent placement
  Interventions: Procedure: Transpancreatic Sphincterotomy

INTERVENTIONS:
Procedure: Needle-Knife Precut Papillotomy over Pancreatic Stent — If the papilla was treated with three unintended MPD cannulations, a needle-knife precut papillotomy with a small incision over a pancreatic stent (NKP-SIPS)
  Arms: NKP-SIPS group
Procedure: Transpancreatic Sphincterotomy — TPS was performed as Goff reported; in short, after cannulation of the pancreatic duct was achieved, a pull-sphincterotome on a guidewire was used to cut the septum between the bile and pancreatic ducts along the direction from 11 o'clock to 12 o'clock. After that, the pancreatic stent is placed first, and the sphincterotomy is extended to expose the biliary lumen, and the biliary duct can be cannulated.
  Arms: TPS group

SUMMARY:
Hello. This study is about a special kind of endoscopy called ERCP, which is used to treat bile duct infections, gallstones, and blockages that cause jaundice. Normally, doctors use a standard method to insert a tube into the bile duct during the procedure. However, even skilled doctors sometimes have trouble - in about 10% to 20% of patients, it's difficult to get the tube in.

When this happens, doctors use advanced techniques called "precut" methods to help make the procedure successful. One of these is called "early needle-knife precut," which is done after trying for 5 minutes without success. Studies have shown this method can reduce the chance of getting pancreatitis (inflammation of the pancreas) afterward.

There are two common types of these advanced techniques:

Needle-knife precut over a pancreatic stent, which gently opens the area using a small cut over a temporary plastic tube.

Transpancreatic sphincterotomy, which also helps open the duct through a different approach.

Both methods can help the procedure succeed and have similar safety results. However, not many studies have compared these two methods early on in the procedure when a pancreatic stent is used.

This study wants to compare them in a safe and scientific way. If you or your family member agrees to join, the doctor will explain everything clearly. Joining is completely voluntary, and saying "no" will not affect the medical care you receive.

DETAILED DESCRIPTION:
Purpose of the Study

This research compares two different advanced techniques used during a special endoscopy procedure (called ERCP) when it is difficult to insert a tube into the bile duct. The goal is to see which method is more successful, takes less time, and causes fewer complications:

Needle-knife precut over a pancreatic stent, and

Transpancreatic sphincterotomy (cutting through the pancreatic opening).

Who Can Join the Study?

Patients may be invited to join this study if they:

Are at least 20 years old

Are receiving their first ERCP treatment

Agree to sign a consent form

Who Cannot Join the Study?

Patients cannot join if they:

Take blood thinners or have bleeding problems

Have tumors causing narrowing in the bile duct or nearby areas

Have certain types of growths near the bile duct opening

Have abnormal intestines from previous surgery

Are currently pregnant

Have active pancreatitis (inflammation of the pancreas)

Have serious infections with symptoms like low blood pressure or difficulty breathing

How the Study Works From November 2021 to October 2023, about 400 patients will be recruited at Kaohsiung Chang Gung Memorial Hospital. If the doctor cannot insert the tube into the bile duct after 5 minutes or if the guidewire enters the pancreatic duct 3 times without success, the patient will be considered to have "difficult cannulation."

Some patients will be placed into groups based on the shape of the bile duct area.

Others will be randomly assigned to one of two groups (like flipping a coin):

Needle-knife precut over a pancreatic stent

Transpancreatic sphincterotomy followed by pancreatic stent placement

Risks and Safety

These procedures are considered safe but can have side effects. Based on past studies:

Pancreatitis (inflammation of the pancreas) may occur in about 6-10% of cases

Bleeding or perforation (a small tear in the intestine) is rare, around 0-2%

Death is very rare, less than 0.5%

Using a pancreatic stent can lower the risk of pancreatitis by about half. However, in very rare cases, the stent might move and require another procedure to remove it.

After the procedure, the patient must not eat or drink until the next day. The medical team will watch for signs of complications such as belly pain, black stool, fever, or confusion. If any of these happen, the doctor will take immediate action. If the patient feels fine the next day, they can slowly begin to eat soft or liquid food.

Joining is Voluntary Participation in the study is completely voluntary. If the patient chooses not to join, it will not affect their regular medical care in any way.

ELIGIBILITY:
Inclusion Criteria:

* At least 20 years old and needed ERCP intervention for obstructive jaundice. They presented the "difficult CBD cannulation".

Exclusion Criteria:

* Patients with successful CBD cannulation within 5 minutes of standard attempts and fewer than three passages of the guidewire into the main pancreatic duct (MPD)
* Previous sphincterotomy,
* Peripapillary diverticula,
* Active pancreatitis,
* Prior gastric surgery,
* Current use of antiplatelet agents,
* Coagulopathy,
* Peri-ampullary tumor-related obstruction,
* Pregnancy,
* Refused or were unable to give informed consent

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-09-28 (Estimated); Study Completion 2025-10-28 (Estimated)

PRIMARY OUTCOMES:
Success rate of common bile duct (CBD) cannulation | During the ERCP procedure (up to 60 minutes)
  Successful selective biliary cannulation using the assigned intervention during the index ERCP session.

SECONDARY OUTCOMES:
Incidence of post-ERCP pancreatitis (PEP) | Within 24 hours after ERCP
  Defined as new or worsened abdominal pain with serum amylase >3 times the upper limit of normal, requiring hospitalization or prolongation of hospital stay.
Incidence of perforation | Within 72 hours after ERCP
  Bleeding categorized as mild (no transfusion), moderate (≤4 units transfused), or severe (≥5 units, angiography, or surgery), with a ≥2 g/dL hemoglobin drop or evidence of melena/hematemesis.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Others, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to concerns regarding patient privacy and institutional policies. In addition, the scope of this single-center study does not include external data sharing in its original ethical approval or informed consent documentation.

REFERENCES:
- [Result] Pecsi D, Farkas N, Hegyi P, Balasko M, Czimmer J, Garami A, Illes A, Mosztbacher D, Par G, Parniczky A, Sarlos P, Szabo I, Szemes K, Szucs A, Vincze A. Transpancreatic sphincterotomy has a higher cannulation success rate than needle-knife precut papillotomy - a meta-analysis. Endoscopy. 2017 Sep;49(9):874-887. doi: 10.1055/s-0043-111717. Epub 2017 Jun 13. PMID 28609791
- [Result] Mariani A, Di Leo M, Giardullo N, Giussani A, Marini M, Buffoli F, Cipolletta L, Radaelli F, Ravelli P, Lombardi G, D'Onofrio V, Macchiarelli R, Iiritano E, Le Grazie M, Pantaleo G, Testoni PA. Early precut sphincterotomy for difficult biliary access to reduce post-ERCP pancreatitis: a randomized trial. Endoscopy. 2016 Jun;48(6):530-5. doi: 10.1055/s-0042-102250. Epub 2016 Mar 18. PMID 26990509

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-09-28): https://cdn.clinicaltrials.gov/large-docs/77/NCT07048977/Prot_SAP_ICF_000.pdf